CLINICAL TRIAL: NCT05704465
Title: Reiki and Qi-gong Therapy Techniques in Improving Negative Emotional States of Anxiety, Depression, and Stress Among Type-2 Diabetic Patients
Brief Title: Reiki and Qi-gong Therapy to Improve Negative Emotional States of Anxiety, Depression, and Stress in Type-2 Diabetics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nagwa Souilm, Assistant Professor of Psychiatric and Mental Health Nursing, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSBS09012023
Record Dates: First submitted 2023-01-09; First posted 2023-01-30 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Type-2 Diabetic Patients
Keywords: Reiki therapy; Qi-gong therapy; Type-2 Diabetic
MeSH Terms: interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki Therapy (Other): Reiki is a biofield therapy technique based on energy healing.
  Interventions: Behavioral: Reiki Therapy
- Qi-gong Therapy (Other): Qigong technique is a type of mind-body meditative exercise developed in traditional Chinese medicine more than 5000 years ago.
  Interventions: Behavioral: Qi-gong Therapy

INTERVENTIONS:
Behavioral: Reiki Therapy — Reiki therapy involved 3 theoretical sessions, 4 practical sessions, and one final one for recapitulation and evaluation. In this technique, energy is guided by therapist's hands placed near patient's body to activate the ability of the body to heal and restore its balance. 1st session for explanation of aim and objectives of program. 2nd one focused on knowledge about negative emotional state. 3rd one discussed Reiki technique and its concept, mode of action, and process. The 4th through 7th sessions were practical. During these sessions, a Reiki practitioner moves his/her hands close to the patient's body in a set of positions. Each hand position focuses on a different part of the body. The hands are held in position for 3 to 10 min., depending on patient's needs. By the end of the session, the patient and therapist reflect on their experience and the emotions with the technique. The eighth session was a recapitulation of the program and ended with evaluation or post-testing.
  Arms: Reiki Therapy
Behavioral: Qi-gong Therapy — Qi-gong involved 3 theoretical sessions, 4 practical sessions, and one final one for recapitulation and evaluation. It involves coordination of breathing and physical movement with mental energy to promote cognitive performance. Both 1st and 2nd sessions were similar to Reiki technique group. The 3rd one addressed the concept of Qi-gong therapy. The 4th through 7th sessions involved patients' doing simple movements and breathing techniques. The practitioner is at about a one-foot distance from the patient's body, to guide and manipulate movements. Breathing patterns are like yoga, with Qigong movements in a mindful link to inspiration and expiration, with incorporation of deep diaphragmatic breathing. The 8th session was similarly for program recapitulation and post-testing.
  Arms: Qi-gong Therapy

SUMMARY:
Diabetes is a worldwide chronic disease due to a disorder in the metabolism of blood glucose. It has high prevalence rates especially in developing countries and is associated with 1.5 million deaths per year. It showed increasing trends over the last few decades. This study aims to To evaluate and compare the effectiveness of Reiki and Qi-gong therapy techniques in improving diabetic patients' negative emotional states. This open-label randomized controlled trial. The study was conducted at the National Institute of Diabetes and Endocrinology's Hospital.

The study sampling population consisted of all patients suffering from Type 2 diabetes attending the setting during the time of the study. randomized into two equal groups: one group will receive reiki intervention, and a second group will receive the qi-gong intervention.

The researcher will use a self-administered questionnaire with a standardized tool (Depression Anxiety Stress Scales [DASS]) for assessment of depression, anxiety, and stress, along with a section for patients' demographic and health characteristics such as age, gender, marital status, duration of diabetes, treatment modalities, body mass index, and glycemic control.

DETAILED DESCRIPTION:
Rationale & background information:

Diabetes is a worldwide chronic disease due to a disorder in the metabolism of blood glucose. It has high prevalence rates especially in developing countries and is associated with 1.5 million deaths per year. It showed increasing trends over the last few decades. Egypt has high prevalence rates of diabetes reaching 20.9% among 20-79 years old, and it ranks tenth highest country in the global ranking of age-adjusted DM prevalence.

Type-1 diabetes mellitus (T1DM) is attributed autoimmune destruction of the β-cells of the pancreas which are responsible for insulin secretion. Meanwhile, in Type-2 diabetes mellitus (T2DM), which is the more prevalent, patients suffer from insulin resistance. These two types are widely different in their etiology, epidemiology, complications, and prognosis although some cases may pose some ambiguity in diagnosis.

Diabetic patients may on the long-term suffer low quality of life due to its physical and psychological complications attributed to macro- and micro-vascular changes leading to renal, retinal, peripheral vascular, cardiovascular, and neurological diseases. Moreover, their risk of death diabetic patients is 1.5 times higher than the general population. Yet, the advances in the treatment modalities of diabetes with the new technologies led to improvements in the life expectancy and prevention of complications among these patients.

In addition to the physical complications associated with Type-2 DM, these patients are at high risk of suffering a wide spectrum of psychological disorders. Thus, diabetic patients are more likely to have negative emotions such as anxiety, depression, and stress. Research has demonstrated high prevalence rates of these psychological problems among diabetic patients. The association between these negative emotion symptoms and diabetes and its trajectory seem to be complicated and bidirectional. For instance, stress and anxiety can increase the risk of developing Type-2 DM through its deregulatory effect on the hypothalamic-pituitary-adrenal axis, thus initiating resistance to insulin. Moreover, depression among was shown to increase the risk of diabetic retinopathy among diabetic patients.

The management of Type-2 DM has greatly evolved during the last few decades, with technological advances reflected on its treatment modalities including self-monitoring, precise insulin titration, and insulin pump, and smart insulin pens. Added to these are the advances in pharmacotherapy, telehealth, and mobile applications.

Complementary and alternative medicine have also added to the effectiveness of treatments of Type-2 DM, and research demonstrated better patient outcomes in multi-approaches compared to mono-approaches in its management. Reflexology, which is based on application of pressure on hands and feet is one of these approaches. Reiki is a biofield therapy technique based on energy healing, developed by the Japanese Mikao Usui of Kyoto in the 19's. In this technique, energy is guided by therapist's hands placed near patient's body to activate the ability of the body to heal and restore its balance. It demonstrated successes in management of fatigue in breast cancer patients on chemotherapy, sleep disorders, hypertension and alcohol consumption, children on palliative care, and cerebral palsy.

Meanwhile, Qigong technique is a type of mind-body meditative exercise developed in traditional Chinese medicine more than 5000 years ago. It involves coordination of breathing and physical movement with mental energy to promote cognitive performance. It showed effectiveness in the management of patients with knee osteoarthritis, atrial fibrillation, pulmonary rehabilitation for COPD, and hypertension.

Significance of the study:

Diabetes mellitus represents a major public health problem in Egypt, with increasing trends. Although recognizing and addressing its related psychological symptoms is of great importance in its management, this still remains suboptimal. Inexpensive complementary medicine approaches like Reiki and Qi-gong therapies could be of help.

Study goals and objectives:

To evaluate and compare the effectiveness of Reiki and Qi-gong therapy techniques in improving diabetic patients' negative emotional states.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes with unchanged antidiabetic therapy Type 2 diabetes with negative emotional state (depression, anxiety, stress)

Exclusion Criteria:

Patients with severe psychiatric Patients with neurological disability or addiction, Patients who unable to perform the intervention techniques Patients who enrolled in other clinical trials were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
effectiveness of Reiki and Qi-gong therapy techniques in improving diabetic patients' negative emotional states. | 8 months
  The response to each statement is on a 4-point scale ranging from "Do not apply to me at all" to "Applies to me very much, or most of the time." These are scored from zero to three, respectively. The total score for each of the three dimensions is computed by simple summation of the scores of its fourteen statements. A higher score of the anxiety dimension denotes that the respondent is apprehensive, shaky, may experience sweating of palms, breathing difficulties, and tachycardia, with possible loss of control

CONTACTS AND LOCATIONS:
Locations (1):
- The National Institute of Diabetes and Endocrinology's Hospital, Cairo, Egypt